CLINICAL TRIAL: NCT00132496
Title: Safety and Efficacy of Rabeprazole in the Treatment of Gastroesophageal Reflux Disease in 12-16 Year Old Patients
Brief Title: Treatment of Gastroesophageal Reflux Disease in 12-16 Year Old Patients With Rabeprazole
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Yufang Lu, Study Director, Eisai Medical Research Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E3810-A001-202
Record Dates: First submitted 2005-08-19; First posted 2005-08-22 (Estimated); Results first posted 2009-12-03 (Estimated); Last update posted 2009-12-03 (Estimated); Status verified 2009-11

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: GERD
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Rabeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: rabeprazole sodium — administered orally and once daily to patients randomized to receive either 10 mg or 20 mg.

SUMMARY:
The primary objective of this study is to collect safety information on rabeprazole 10 mg and 20 mg in the treatment of gastroesophageal reflux disease (GERD) in children aged 12 to 16 years. The secondary objectives are to assess the efficacy of rabeprazole on the improvement of the symptoms of GERD and to explore the relationship of symptom relief to dose received, based on symptom frequency and severity, antacid use, and quality of life (QOL) measures.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged 12 to 16 years with a clinical diagnosis of symptomatic GERD or suspected or endoscopically proven GERD.
2. Patients who have ever been treated with, or are currently receiving proton pump inhibitors (PPIs),histamine receptor (H2) blockers, or antacids are eligible (as long as they can go off PPIs and H2 blockers for three days prior to dosing, except for cimetidine, which must be discontinued for at least seven days prior to dosing; exclusion criteria 5 and 6). Also, patients should be able to go off PPI therapy for two weeks at the end active drug treatment.
3. Children with stable asthma/reactive airways disease on stable treatment regimens are eligible.
4. Children on stable doses of allergy, antiepileptic, antidepressant, and attention deficit disorder medicines are eligible.
5. Patients must be able and willing to swallow the test drug tablet intact. The ability of the child to swallow an intact tablet must be confirmed by the site at Screening.
6. The patient is willing and able to give assent to participate.
7. The patient's parent or guardian gives written informed consent.
8. Post-pubertal females will be required to be abstinent during the course of the study.
9. Clinically insignificant laboratory findings.

Exclusion Criteria:

1. Evidence of significant hepatic, renal, respiratory, endocrine, immune, infectious, hematologic, neurologic, psychiatric, or cardiovascular system abnormalities that would interfere with the conduct of the study, the interpretation of study results, or the health of the patient during the study.
2. History of primary esophageal motility disorders or systemic condition affecting the esophagus (eg, scleroderma, esophageal infections).
3. History of eosinophilic esophagitis, persistent milk protein allergy, or allergic gastroenteropathy. History or current presence of peptic ulcers; current presence of Helicobacter pylori.
4. History of definitive acid-lowering surgery, previous esophageal surgery, or esophageal stricture is disallowed. History of fundoplication or feeding tube insertion is allowed.
5. Treatment with full therapeutic doses of H2-receptor antagonists or sucralfate within three days prior to dosing (or a shorter washout if agreed to by Investigator and Sponsor), except for cimetidine, which must be discontinued for at least seven days prior to dosing.
6. Treatment with a proton pump inhibitor within three days prior to dosing (or a shorter washout if agreed to by Investigator and Sponsor).
7. Inability to have 2-week PPI therapy-free period at end of active drug treatment.
8. Pregnancy or lactation.
9. Known or suspected drug addiction or alcohol abuse and/or a positive urine drug screen not explained by medication list; occasional alcohol or tobacco use is not an exclusion criterion.
10. Unwilling or unable to abide by the requirements of the study or violating the prohibitions and restrictions of the study defined in Section 9.4.
11. Any condition which would make the patient, in the opinion of the Investigator or Sponsor, unsuitable for the study.
12. Participation in another investigational drug study within one month prior to dosing.
13. A history of allergy/sensitivity to proton pump inhibitors or to their inactive ingredients.

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 111 (Actual)
Dates: Start 2005-08; Primary Completion 2006-05 (Actual); Study Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yufang Lu, Study Director — Eisai Inc.
Locations (25):
- United States (25):
  - Longmont Medical Research Network, Longmont, Colorado
  - Nova Southeastern University, Fort Lauderdale, Florida
  - Babies and Beyond Peds, New Port Richey, Florida
  - Dr. Patricia Barrington, Dr. B. Abraham, PC, Snellville, Georgia
  - Multi-specialty Clinical Research, Hoffman Estates, Illinois
  - Kentucky Pediatric/Adult Research, Bardstown, Kentucky
  - Professional Clinical Research, Cadillac, Michigan
  - Community Pediatric Associates, Kalamazoo, Michigan
  - The Center for Human Nutrition, Omaha, Nebraska
  - Children's Hospital of Buffalo - Digestive Disease And Nutrition Center, Buffalo, New York
  - Winthrop University Hospital, Mineola, New York
  - Pediatric Associates of Mount Carmel, Inc., Cincinnati, Ohio
  - Pediatric Associates of Mt. Carmel, Cincinnati, Ohio
  - University of Pediatrics, Mason, Ohio
  - Center for Children's Digestive Health, Youngstown, Ohio
  - Pharmacotherapy Research Associates, Zanesville, Ohio
  - Biomedical Research Associates, Shippensburg, Pennsylvania
  - DeGarmo Institute of Medicine Research, Greer, South Carolina
  - Focus Research Group, Hendersonville, Tennessee
  - ProMed Healthcare, Johnson City, Tennessee
  - NE Ohio University College of Medicine, Lebanon, Tennessee
  - Southwest Children's Research Associates, San Antonio, Texas
  - Alpine Medical Group, Salt Lake City, Utah
  - Rockwood Clinic North, Spokane, Washington
  - Marshall University, Huntington, West Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was recruited at 25 centers in the US during the period of 18-Aug-2005 and 1-May-2006.
Pre-assignment Details: There was a screening period of up to 2 days before treatment assignment
Groups:
- Rabeprazole 10 mg; Rabeprazole 20 mg: once daily for 8 weeks
Period: Overall Study
Arm/Group | Rabeprazole 10 mg | Rabeprazole 20 mg
Started | 54 | 57
Completed | 52 | 55
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rabeprazole 10 mg | Rabeprazole 20 mg | Total
Number analyzed (Participants) | 54 | 57 | 111
Age Continuous [Mean (Standard Deviation); unit: years] | 14.2 (1.3) | 14.1 (1.5) | 14.2 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 26 | 53
  Male | 27 | 31 | 58
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 0 | 0 | 0
  Black or African American | 4 | 1 | 5
  White | 47 | 53 | 100
  Hispanic | 1 | 2 | 3
  Other | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 54 | 57 | 111

OUTCOME MEASURES:

1. Primary Outcome: Treatment-emergent Adverse Events Experienced by >=5% of Patients in Any Treatment Group
Description: Primary safety outcomes include adverse events, physical examinations and clinical laboratory results. AE results are presented in the table.
Time Frame: 8 weeks from randomization and end of treatment
Population: Safety population (all patients who received at least one dose of study treatment) was the primary analysis population.
Measure: Number; unit: Participants
Arm/Group | Rabeprazole 10 mg | Rabeprazole 20 mg
Number analyzed (Participants) | 54 | 57
Participants
  Diarrhea | 3 | 2
  Nausea | 3 | 2
  Upper abdominal pain | 1 | 3
  Chest pain | 0 | 3
  Upper respiratory tract infection | 4 | 3
  Bronchitis | 3 | 2
  Pharyngitis | 3 | 2
  Sinusitis | 2 | 3
  Nasopharyngitis | 1 | 4
  Otitis media | 1 | 3
  Headache | 5 | 6
  Pharyngolaryngeal pain | 6 | 5
  Cough | 5 | 3
  Nasal congestion | 4 | 4
  Total # subjects reporting AEs | 41 | 45

ADVERSE EVENTS:
Arm/Group | Rabeprazole 10 mg | Rabeprazole 20 mg
Serious Adverse Events (participants affected / at risk) | 0 | 1
Other Adverse Events (participants affected / at risk) | 41 | 45
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Rabeprazole 10 mg | Rabeprazole 20 mg
Mood swings (Nervous system disorders) | 0/54 (0) | 1/57 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Rabeprazole 10 mg | Rabeprazole 20 mg
Diarrhea (Gastrointestinal disorders) | 3/54 | 2/57
Nausea (Gastrointestinal disorders) | 3/54 | 2/57
Upper andominal pain (Gastrointestinal disorders) | 1/54 | 3/57
Chest Pain (General disorders) | 0/54 | 3/57
Upper respiratory tract infection (Infections and infestations) | 4/54 | 3/57
Bronchitis (Infections and infestations) | 3/54 | 2/57
Pharyngitis (Infections and infestations) | 3/54 | 2/57
Sinusitis (Infections and infestations) | 2/54 | 3/57
Nasopharyngitis (Infections and infestations) | 1/54 | 4/57
Otitis media (Infections and infestations) | 1/54 | 3/57
Headache (Nervous system disorders) | 5/54 | 6/57
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 6/54 | 5/57
Cough (Respiratory, thoracic and mediastinal disorders) | 5/54 | 3/57
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4/54 | 4/57

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other